CLINICAL TRIAL: NCT04800094
Title: Pilot Study of On-Cart Liver Fat Quantification (LFQ) Feature to Assess Correlation With Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) Results in a Pediatric Population
Brief Title: Pediatric Liver Fat Quantification (LFQ) Phase 2 Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-GIS-10983
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2024-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis
Keywords: Liver Fat Quantification; Ultrasound; Liver Disease; Digestive System Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Digestive System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Investigational Ultrasound Imaging for Liver Fat Quantification (Experimental)
  Interventions: Device: Investigational Liver Fat Quantification Software

INTERVENTIONS:
Device: Investigational Liver Fat Quantification Software — All subjects enrolled in this study will undergo two abdominal ultrasound examinations using the investigational Liver Fat Quantification feature on the Philips EPIQ Ultrasound System. In addition, all subjects will also undergo one MRI-PDFF examination according to the clinical standard of care.

SUMMARY:
This clinical study will involve performing a series of medical imaging procedures of the abdomen using both ultrasound and MRI modalities in subjects at risk for or already diagnosed with Nonalcoholic Fatty Liver Disease (NAFLD). The primary objective of this clinical study is to evaluate the clinical feasibility of an investigational ultrasound technique for quantifying liver fat by comparing specific ultrasound-derived biomarkers with the liver fat percentage obtained from MRI Proton Density Fat Fraction (MRI-PDFF) measurements. All subjects enrolled in this study will undergo one investigational abdominal ultrasound examination using the Philips EPIQ Ultrasound System and one MRI PDFF examination according to the clinical standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 5 years old up through and including 21 years old who are able to provide informed consent to participate or have a legal representative/parent/legal guardian who is able to provide informed consent for the subject to participate.
* Subjects must be eligible for a standard abdominal ultrasound examination and standard non-contrast MRI examination.

In addition, at least one of the following criteria must also be met:

* Overweight or obese (BMI-for-age ≥ 85th percentile).
* Diagnosed with Type 2 diabetes per standard clinical guidelines.
* Diagnosed with hypercholesterolemia per standard clinical guidelines.
* Diagnosed with or clinically suspected of having NAFLD/NASH based on previous medical record, medical imaging, liver biopsy, and/or laboratory testing.

Exclusion Criteria:

* History of moderate/heavy/binge alcohol consumption exceeding NIAAA guidelines.
* Evidence of hepatotoxicity or cirrhosis in the clinical judgment of the investigator.
* History of chronic liver disease other than NAFLD (e.g., viral, cholestatic, or autoimmune).
* Use of drugs associated with hepatic steatosis:

  * Amiodarone
  * Methotrexate
  * Nucleoside reverse transcriptase inhibitors (didanosine, stavudine)
  * Valproic acid
  * Dexamethasone
  * Tamoxifen
  * 5-FU-based adjuvant chemotherapy
  * Apo-B inhibitors (mipomersen, lomitapide)
  * Tetracycline exceeding 2 g/day
  * Acetylsalicylic acid exceeding 150 mg/kg

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smita S Bailey, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 10
Weight [Mean (Standard Deviation); unit: kg] | 67.9 (126.5)
Height [Mean (Standard Deviation); unit: cm] | 151.3 (16.5)

OUTCOME MEASURES:

1. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements of Hepatorenal Index (HRI) Ultrasound Biomarker for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. The difference between the two operators was calculated at the subject level by averaging multiple measurements. To assess the correlation between measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 60 non missing scans reviewed for this study. The primary outcome measure, the Hepatorenal Index, was calculated based on these scans. The hepatorenal index measurement from each ultrasound scan was reviewed.
Measure: Mean (Standard Deviation); unit: Hepatorenal Index
Units Other Than Participants: Ultrasound scans
Groups:
- Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification: Investigational Liver Fat Quantification Software: All subjects enrolled in this study will undergo two abdominal ultrasound examinations using the investigational Liver Fat Quantification feature on the Philips EPIQ Ultrasound System. In addition, all subjects will also undergo one MRI-PDFF examination according to the clinical standard of care.
Arm/Group | Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Number analyzed (Ultrasound scans) | 60
Hepatorenal Index | 1.7 (0.7)
Statistical Analysis 1: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Hepatorenal Index (HRI)" derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome; Test type: Other — Pearson correlation coefficient was calculated based on all measurements assuming independency; Pearson correlation coefficient = 0.4459
Statistical Analysis 2: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 1, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject level averages of multiple measurements; Pearson correlation coefficient = 0.5431
Statistical Analysis 3: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 1, analysis 1]; Test type: Other — To account for within subject variance in repeated measures by two different operators, a method with MIXED model for repeated measurements was used to estimate the correlation between two techniques with repeated measures. An unstructured covariance matrix was used; Mixed Model = 0.4871

2. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements of Acoustic Attenuation (dB/cm/MHZ) Ultrasound Biomarker for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. To assess the correlation between subject averaged measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record.
  Correlation of each ultrasound biomarker with the liver fat percentage reported from MRI-PDFF is assessed independently to evaluate individual biomarker performance. A higher attenuation value indicates worse liver condition, while a lower attenuation value suggests better liver status.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 60 scans reviewed for this study. The primary outcome measure, the Acoustic Attenuation (dB/cm/MHZ), was evaluated based on these scans. The acoustic attenuation from each ultrasound was reviewed.
Measure: Mean (Standard Deviation); unit: dB/CM/MHz
Units Other Than Participants: ultrasound scans
Groups:
- Acoustic Attenuation: Investigational Ultrasound Imaging for Liver Fat Quantification: Investigational Liver Fat Quantification Software: All subjects enrolled in this study will undergo two abdominal ultrasound examinations using the investigational Liver Fat Quantification feature on the Philips EPIQ Ultrasound System. In addition, all subjects will also undergo one MRI-PDFF examination according to the clinical standard of care.
Arm/Group | Acoustic Attenuation: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Number analyzed (ultrasound scans) | 60
dB/CM/MHz | 0.6 (0.1)
Statistical Analysis 1: Comparison: Acoustic Attenuation: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Acoustic attenuation " derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record; Test type: Other — Pearson correlation coefficient was calculated based on all measurements assuming independency; Pearson correlation coefficient = 0.1742
Statistical Analysis 2: Comparison: Acoustic Attenuation: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 2, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject averages of multiple measurements; Pearson correlation coefficient = 0.1770
Statistical Analysis 3: Comparison: Acoustic Attenuation: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; Correlation estimated from a mixed model = 0.1756

3. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements of Tissue Stiffness (kPa) Ultrasound Biomarkers for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. To assess the correlation between subject averaged measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record. This measured the MRI PDFF fat fraction used as the standard to evaluate the Tissue stiffness (kPa) measurements.
  Correlation of each ultrasound biomarker with the liver fat percentage reported from MRI-PDFF is assessed independently to evaluate individual biomarker performance.
  Correlation of each ultrasound biomarker with the liver fat percentage reported from MRI-PDFF will be assessed independently to evaluate individual biomarker performance.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 60 scans reviewed for this study. Two scans were not usable and were excluded from the analysis. So, a total of 58 scans were included for this analysis.
Measure: Mean (Standard Deviation); unit: kPa
Units Other Than Participants: Ultrasound scans
Groups:
- Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification: Investigational Liver Fat Quantification Software: All subjects enrolled in this study will undergo two abdominal ultrasound examinations using the investigational Liver Fat Quantification feature on the Philips EPIQ Ultrasound System. In addition, all subjects will also undergo one MRI-PDFF examination according to the clinical standard of care.
Arm/Group | Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Number analyzed (Ultrasound scans) | 58
kPa | 6.6 (1.6)
Statistical Analysis 1: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Tissue stiffness" derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record; Test type: Other — Pearson correlation coefficient was calculated based on all observations assuming independency; Pearson correlation coefficient = 0.0810
Statistical Analysis 2: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 3, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject averages of multiple measurements; Pearson correlation coefficient = 0.0902
Statistical Analysis 3: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; Correlation estimated from a mixed model = 0.0841

4. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker "Hepatorenal Index (HRI)"
Description: To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition. The difference between the two operators was calculated at the subject level by averaging multiple measurements. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome.
Time Frame: Intra-procedural (1 day)
Population: The analysis included 60 ultrasound scans, performed by two different operators, from 30 enrolled participants. The hepatorenal index measurement was calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: Hepatorenal Index
Units Other Than Participants: Ultrasound scans
Arm/Group | Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Number analyzed (Ultrasound scans) | 60
Hepatorenal Index | -0.5 (0.6)
Statistical Analysis 1: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to test the same day inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.36, 95% CI 2-sided [0.02 to 0.63]

5. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker "Hepatorenal Index (HRI)"
Description: To evaluate the LFQ data acquisition failure rate, the proportion of subjects who have at least one unacceptable image quality due to inadequate acoustic scanning windows, motion artifacts, or other technical limitations
Time Frame: Intra-procedural (1 day)
Population: To quantify the number of overall subjects with at least one unacceptable image quality
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Participants | 0
Statistical Analysis 1: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Hepatorenal Index (HRI)"; Test type: Other — The proportion of subjects who have at least one unacceptable image quality due to inadequate acoustic scanning windows, motion artifacts, or other technical limitations and the associated 2-sided 95% binomial confidence intervals were calculated and summarized by each operator and overall; Proportion = 0, 95% CI 2-sided [0 to 0]

6. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker Acoustic Attenuation (dB/cm/MHZ)
Description: To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition.
  The difference between the two operators was calculated at the subject level by averaging multiple measurements.
Time Frame: Intra-procedural (1 day)
Population: The analysis included 60 ultrasound scans, performed by two different operators, from 30 enrolled participants. The acoustic attenuation (dB/cm/MHZ) measurement was calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: dB/cm/MHZ
Units Other Than Participants: ultrasound scans
Arm/Group | Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Number analyzed (ultrasound scans) | 60
dB/cm/MHZ | -0.01 (0.02)
Statistical Analysis 1: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the difference in quantitative ultrasound biomarker Acoustic attenuation measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to assess the same day inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.94, 95% CI 2-sided [0.88 to 0.97]

7. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker Tissue Stiffness (kPa)
Description: as for outcome 6
Time Frame: Intra-procedural (1 day)
Population: The analysis included 58 ultrasound scans, performed by two different operators, from 29 enrolled participants. The Tissue stiffness (kPa) measurement was calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: Tissue stiffness (kPa)
Units Other Than Participants: ultrasound scans
Arm/Group | Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 29
Number analyzed (ultrasound scans) | 58
Tissue stiffness (kPa) | 0.7 (1.2)
Statistical Analysis 1: Comparison: Hepatorenal Index: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 4, analysis 1]; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to test the inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.63, 95% CI 2-sided [0.36 to 0.8]

8. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker Tissue Stiffness (kPa)
Description: as for outcome 5
Time Frame: Intra-procedural (1 day)
Population: 30 participants enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Participants | 2
Statistical Analysis 1: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Tissue stiffness (kPa)"; Test type: Other — [test comment as in outcome 5, analysis 1]; Proportion = 6.7, 95% CI 2-sided [0.0 to 15.6]

9. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker Acoustic Attenuation (dB/cm/MHZ)
Description: as for outcome 5
Time Frame: Intra-procedural (1 day)
Population: 30 participants enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 30
Participants | 0
Statistical Analysis 1: Comparison: Tissue Stiffness: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Acoustic attenuation (dB/cm/MHZ)"; Test type: Other — [test comment as in outcome 5, analysis 1]; Proportion = 0, 95% CI 2-sided [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Up to 8 weeks from enrollment to completion of all study-related procedures
Description: No significant foreseeable safety events are associated with this study. No significant ADEs are anticipated because the study procedure is limited to noninvasive diagnostic ultrasound imaging using the investigational LFQ software. The Philips EPIQ Ultrasound System with investigational LFQ software and probes comply with harmonized safety standards governing all diagnostic ultrasound imaging devices and pose no additional risk beyond that associated with any other ultrasound imaging procedure
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT04800094/Prot_SAP_000.pdf